CLINICAL TRIAL: NCT07234513
Title: Diabetes Mellitus Symptoms Related to Physical Competence: Do They Predict Dynamic Balance?
Brief Title: Diabetes Mellitus Symptoms Related to Physical Competence
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Mehmet Duray, Assoc. Prof., Suleyman Demirel University
Other Study IDs: 60116787-020/71477
Record Dates: First submitted 2025-09-23; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Dynamic Balance; Physical Activity; Exertion; Urinary Incontinence
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: There will be only one group in the study.
  Interventions: Diagnostic Test: There will be no intervention in the study. Only descriptive tests will be used.

INTERVENTIONS:
Diagnostic Test: There will be no intervention in the study. Only descriptive tests will be used. — There will be no intervention in the study. Only descriptive tests will be used.

SUMMARY:
The research is a cross-sectional study and was planned to determine which diabetes mellitus symptoms related to physical competence have a greater impact on balance in patients with diabetes mellitus

DETAILED DESCRIPTION:
The present study was designed as a cross-sectional observational study to investigate the relationship between diabetes mellitus (DM)-related symptoms and physical competence, with a specific focus on balance performance in individuals diagnosed with DM. Considering that diabetes is a chronic metabolic disease that frequently leads to multisystemic complications such as peripheral neuropathy, muscle weakness, sensory impairments, and reduced physical capacity, it is essential to determine how these clinical manifestations affect functional outcomes. Since balance is a critical component of daily living activities and directly influences fall risk, mobility, and quality of life, identifying which DM-related symptoms most strongly contribute to balance impairment may provide important insights for rehabilitation and preventive strategies. By assessing symptom domains related to physical competence and their association with balance performance, this study aims to reveal the key determinants of postural control in patients with DM, thereby guiding both clinical evaluation and individualized intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* having Diabetes MEllitus
* having a Mini Mental Test (MMT) score ≥ 24

Exclusion Criteria:

* the presence of comorbid conditions that could affect balance, such as lower extremity injuries, musculoskeletal surgery, diabetic neuropathy, orthopedic, neurological and cardiovascular diseases, and hearing or vision problems.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Diabetes Mellitus
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-07-13 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | 7 months
  Four-Step Square Test (FSST): Two strips were placed perpendicular to each other on the floor to create 4 squares. At the start of the test, the patient stood on square 1 facing square 2. The stepping sequence was as follows: 2-3-4-1-4-3-2-1. Participants were instructed to complete the sequence as fast as possible, without touching the canes or strips, and to ensure that both feet fully contacted the ground in each square. If the participant failed to complete the sequence correctly, lost balance, or touched the cane, the test was repeated. The total time required to complete the test was recorded

SECONDARY OUTCOMES:
International Physical Activity Questionnaire-Long Form (IPAQ-LF) | 7 months
  The IPAQ-LF consists of 27 items designed to assess physical activity across various domains, such as of housework, gardening, work activities, transportation, and leisure activities. The weekly physical activity level was calculated as metabolic equivalent of task (MET), by multiplying the activity duration in the previous week. An increase in the score indicates a high level of physical activity. According to the results, participants can be classified as inactive, minimally active, or very active.
  Inactive (Category 1): The lowest level of physical activity. Situations that do not meet the criteria for Categories 2 or 3 are considered "inactive."
  Minimally Active (Category 2): Achieving a minimum of 600 MET-min/week, with vigorous activity performed for at least 20 minutes per day on 3 or more days.
  Very Active (Category 3): At least 3 days of vigorous activity achieving a minimum of 1500 MET-min/week.
6-Minute Walking Test (6MWT) | 7 months
  6-Minute Walking Test (6MWT): The 6MWT is a valid, reliable, and gold standard maximal exercise effort test, that evaluates functional capacity and aerobic efficiency. The 6MWT was performed between two cones placed 30 m apart. Before the test, the physiotherapist recorded the vital signs (blood pressure, heart rate and respiratory rate per minute). The participants were asked to walk as fast as possible for 6 min and were informed in the last 1 min. If the patient had to stop walking within 6 min, they were asked to lean against the wall, but no patient stopped walking. The assessments were repeated at the end of the 6MWT, and the walking distance was recorded in meters.
Modified Borg Scale (MBS) | 7 months
  Modified Borg Scale (MBS): The MBS is a modified version of the Borg Rating of Perceived Exertion Scale, which was developed to quantify the subjective level of effort experienced during physical activity. The scale is commonly used in clinical rehabilitation to quantify the rates of fatigue-related perceived exertion between 0 and 10. "0" equates to "at rest" and "10" equates to "very, very hard".
International Urinary Incontinence Consultation Questionnaire-Short Form (ICIQ-UI SF) | 7 months
  International Urinary Incontinence Consultation Questionnaire-Short Form (ICIQ-UI SF): The ICIQ-UI SF, consisting of 6 items questioning the frequency, amount, and duration of urinary incontinence, and the impact of these complaints on daily life. The ICIQ-UI SF, is a short and simple questionnaire, that is useful in screening incontinence and obtaining brief but comprehensive data on the level, impact, and perceived effects of incontinence symptoms. The highest possible score on the questionnaire is 21. A higher score indicates a greater impact of incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: ÇETİŞLİ KORKMAZ, Study Director — Pamukkale University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT07234513/Prot_SAP_000.pdf